CLINICAL TRIAL: NCT03309774
Title: Complex Regional Pain Syndrome in Children: Impact of Bergès Relaxation on the Autonomic Balance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failing of recruitment
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1708124; 2017-A02092-51 (Other: ANSM)
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: Children; Complex Regional Pain Syndrome; Relaxation; Bergès relaxation; Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complex Regional Pain Syndrome (CRPS) (Experimental): Children 6 to 12 years old child with Complex Regional Pain Syndrome (CRPS) type 1 will be included.
  They will have questionnaires, holter electrocardiogram, blood pressure and relaxation sessions.
  Interventions: Diagnostic Test: questionnaires; Diagnostic Test: holter electrocardiogram; Diagnostic Test: blood pressure; Other: relaxation sessions

INTERVENTIONS:
Diagnostic Test: questionnaires — Children with Complex Regional Pain Syndrome (CRPS) will be filled questionnaires before and after relaxation sessions. These questionnaire evaluate the quality of life and pain of child
  There will be:
  * Questionnaire KIDSCREEN 52
  * Visual Analogue Scale (EVA)
  * Neuropathic Pain 4 (DN4)
  * Pain of the child Gustave Roussy (DEGR)
Diagnostic Test: holter electrocardiogram — Children with Complex Regional Pain Syndrome (CRPS) will be have holter electrocardiogram before and after relaxation sessions.
Diagnostic Test: blood pressure — Blood pressure of Children with Complex Regional Pain Syndrome (CRPS) will be measured by Nexfin monitor before and after relaxation sessions.
Other: relaxation sessions — Children with Complex Regional Pain Syndrome (CRPS) will be performed 20 relaxation sessions and 2 per week.
  During relaxation sessions children will be recorded by voice recorder. Children should describe his feelings at the preceding session.
  After every relaxation sessions children evaluate pain according to Eland Color Scale.

SUMMARY:
Complex regional pain syndrome (CRPS) is a disease provoking chronic pain in the limbs, following a trauma. Patient care is complicated by the variable clinical picture and response to treatment. The stress level of the organization, for chronic pain impacts the regulation of the autonomic balance. The study of time and frequency domain analysis of Heart Rate Variability (HRV) allows non-invasive and reproducible assessment of the autonomic balance.

DETAILED DESCRIPTION:
The hypothesis in this study is that the sympathovagal balance could be altered in children with CRPS. But the impact of relaxation on pain and balance has been proven. This study aims to assess the impact of the assumption by the relaxation therapy in children suffering from CRPS, on sympathovagal balance.

It is an experimental prospective single-center study to highlight after a standardized relaxation program, changes in the time and frequency indices variability in heart rate, parameters of pain and quality of life with the CRPS children 6 to 16 years.

ELIGIBILITY:
Inclusion Criteria:

* Parents affiliates or entitled to a social security scheme
* Children from 6 to 16 years with Complex Regional Pain Syndrome (CRPS) type 1
* Diagnosis according to the Budapest criteria.

Exclusion Criteria:

* Child with pathologies reaching the central nervous system or the brain stem.
* Children with a severe pathology of cardio-respiratory or heart being referred to treatment.
* Children requiring emergency surgery or trauma or septic or inflammatory context.
* Children with some psychiatric diseases
* Children who no understand french enough

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
high frequency index | at 3 months
  measured by holter electrocardiogram.

SECONDARY OUTCOMES:
blood pressure | at 3 months
life quality of children | at 3 months
  by questionnaire KIDSCREEN 52
evaluation of pain | at 3 months
  by questionnaire EVA
evaluation of pain | at 3 months
  by questionnaire DN4
evaluation of pain | at 3 months
  by questionnaire DEGR
intensity of pain | at 3 months
  with Eland Color Scale
location of pain | at 3 months
  with Eland Color Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gautheron, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No